CLINICAL TRIAL: NCT02833051
Title: The Impact of an Acute Bout of Exercise on Children's Eating Behaviors
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Assistant Professor, Penn State University
Other Study IDs: EnergyBalance01
Record Dates: First submitted 2016-06-08; First posted 2016-07-14 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to examine the effects of an acute bout of exercise on children's energy intake over the course of a day. Previous studies in adolescents and adults have shown exercise to be effective in decreasing short-term energy intake, with some variability. Individual characteristics such as habitual physical activity and psychological factors may influence the effect of exercise on energy intake, but these factors have yet to be examined. The investigators have assembled a multi-disciplinary team of researchers, with expertise in eating behavior, exercise, psychology, and clinical research in order to examine these questions. First, the investigators will examine the difference in energy intake at lunch, snack, and dinner meals in response to 30 minutes of imposed exercise compared to 30 minutes of rest. Second, the investigators will collect objective measures of children's habitual physical activity, child characteristics (body composition, eating behavior traits), and individual responses to the controlled exercise bout. The investigators can then examine both group and individual differences in the energy intake response to exercise. Children (ages 9-12) will be tested over the course of three visits. The key outcome will be differences in energy intake in response to exercise vs. rest. Secondary outcomes include the influence of differences in habitual physical activity, personal characteristics, and responses to the exercise bout on children's energy intake. The long term goal of this line of research is to understand the mechanisms behind the interaction between exercise and energy intake. The translational potential of this research will be to inform personalized childhood obesity prevention strategies in children at risk for overweight.

ELIGIBILITY:
Inclusion Criteria:

* English as a native language
* Reading at/above grade level
* Generally healthy
* Child is "normal weight" below the 85% age- and sex-specific BMI percentile
* Child has at least one biological parent classified as "overweight" or "obese" (≥ 25 kg/m^2)
* Regularly eats breakfast

Exclusion Criteria:

* Contraindications to exercise testing (as defined by the American College of Sports Medicine)
* Medical conditions
* Psychiatric conditions
* Participation in competitive sports teams (year-round or more than 3 practices / week)
* Food allergies or other dietary restrictions

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 9-12 years old
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Baseline energy intake | Collected at week 1 of the study
  Food intake is measured at objective laboratory test-meals as the difference between the pre-meal and post-meal weights of individual food items served. Weight of food is converted to energy in kilocalories based on nutrition facts label information.
Energy intake following exercise | Collected at week 2 or 3 (randomized) of the study
  Food intake is measured at objective laboratory test-meals as the difference between the pre-meal and post-meal weights of individual food items served. Weight of food is converted to energy in kilocalories based on nutrition facts label information.
Energy intake following sedentary control | Collected at week 2 or 3 (randomized) of the study
  Food intake is measured at objective laboratory test-meals as the difference between the pre-meal and post-meal weights of individual food items served. Weight of food is converted to energy in kilocalories based on nutrition facts label information.
Activity-related energy expenditure - Baseline day | Collected in the laboratory at week 1, 2, and 3, and at home for one week between the 2nd and 3rd laboratory visits
  Measured using ActiGraph accelerometers
Activity-related energy expenditure - Exercise day | Collected at week 2 or 3 (randomized) of the study
  Measured using ActiGraph accelerometers
Activity-related energy expenditure - Sedentary control day | Collected at week 2 or 3 (randomized) of the study
  Measured using ActiGraph accelerometers

SECONDARY OUTCOMES:
Baseline submaximal fitness test performance | Collected at week 1 of the study
  YMCA submaximal cycle ergometer test - American College of Sports Medicine
Exercise test performance (70% intensity) - Heart rate | Collected at week 2 or 3 (randomized) of the study
  Measured by Polar Heart Rate Monitor
Exercise test performance (70% intensity) - Blood pressure | Collected at week 2 or 3 (randomized) of the study
  Measured by registered nurse or trained research assistant
Exercise test performance (70% intensity) - Ratings of perceived exertion | Collected at week 2 or 3 (randomized) of the study
  Measured on the Borg Scale
Exercise test performance (70% intensity) - Completion | Collected at week 2 or 3 (randomized) of the study
  Children's completion of the full 30 minutes of 70% intensity exercise
Child sleep patterns | Collected at home for one week between the 2nd and 3rd laboratory visits
  Measured using ActiGraph accelerometers
Child physical activity patterns | Collected at home for one week between the 2nd and 3rd laboratory visits
  Measured using ActiGraph accelerometers

OTHER OUTCOMES:
Liking of foods | Collected at week 1 and 2 of the study
  Ratings of how much child likes specific foods used in the study test meals, completed on visual analog scales
Wanting of foods | Collected at week 1 and 2 of the study
  Ratings of how much child wants to eat specific foods used in the study test meals, completed on visual analog scales
Fullness feelings | Collected at multiple time points during weeks 1, 2, and 3
  Ratings of how full the child feels on a child friendly visual analog scale
Height | Collected at week 1
  Height in cm measured by stadiometer
Weight | Collected at week 1
  Weight in kg by standard digital scale
Body fat percentage | Collected at week 1
  Assessed by bioelectrical impedance analysis scale
Body mass index | Collected at week 1
  Calculated from height and weight (kg/m^2)
BMI percentile | Collected at week 1
  Calculated from height, weight, age, sex
BMI z-score | Collected at week 1
  Calculated from height, weight, age, sex
Fat mass index | Collected at week 1
  Calculated from body fat percentage, weight, height
Fat-free mass index | Collected at week 1
  Calculated from fat mass, weight, height
Appetitive traits | Collected at week 1
  Parent-reported questionnaire of habitual eating styles in children
Pubertal development | Collected at week 1
  Parent-reported questionnaire
Family demographics | Collected at week 1
  Parent-reported questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No